CLINICAL TRIAL: NCT00004408
Title: Phase III Randomized Study of Poloxamer 188 for Vaso-Occlusive Crisis of Sickle Cell Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Collaborators: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13296; CYTRX-C97-1248; CYTRX-FDR001433
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Sickle Cell Anemia
Keywords: disease-related problem/condition; genetic diseases and dysmorphic syndromes; hematologic disorders; pain; rare disease; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Genetic Diseases, Inborn; Hematologic Diseases; Pain; Rare Diseases | interventions — Poloxamer

INTERVENTIONS:
Drug: poloxamer 188

SUMMARY:
OBJECTIVES: I. Assess the efficacy of poloxamer 188 in reducing the duration of painful vaso-occlusive crisis in patients with sickle cell disease.

II. Assess the effect of poloxamer 188 on duration and intensity of pain, total analgesic use, and length of hospitalization of these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to hydroxyurea use.

Patients are randomized to treatment poloxamer 188 or placebo. Treatment begins within 12 hours of presentation with crisis. Patients receive poloxamer 188 or placebo by continuous infusion for 48 hours. Pain is assessed before, during, and after treatment.

Patients are followed on days 7-14 and 28-35.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Sickle cell disease confirmed by electrophoresis or high pressure liquid chromatography
* At least one prior documented painful crisis episode but no greater than 10 crises per year for the last two years
* Sudden onset of acute pain lasting 4-12 hours and involving at least one site
* Severe crisis pain that requires parenteral analgesics and hospitalization, but not within the preceding 2 weeks

--Prior/Concurrent Therapy--

* Surgery: At least 2 weeks since prior major surgery No concurrent surgery
* Other: At least 2 weeks since prior puncture of noncompressible vessels No prior therapy using poloxamer 188 No concurrent investigational drug No concurrent use of nonsteroidal anti-inflammatory drugs

--Patient Characteristics--

* Hematopoietic: No significant bleeding or bleeding disorder
* Hepatic: ALT no greater than 2 times normal
* Renal: No active renal disease Creatinine no greater than 1.0 mg/dL OR Creatinine clearance greater than 50 mL/min Protein less than 300 mg/dL
* Cardiovascular: No evidence of acute myocardial ischemia or infarction
* Neurologic: At least 6 months since prior cerebrovascular accident or seizure
* Other: Not pregnant Fertile patients must use effective contraception during and for at least 30 days after treatment No history of chronic bacterial osteomyelitis No history of drug or alcohol abuse At least 6 months since prior use of illicit drug Have adequate IV access No crisis with life-threatening complications such as: Hepatic or splenic sequestration Acute chest syndrome Aplastic crisis No known infection or infection with encapsulated organism No evidence of septic shock Not concurrently hospitalized for other conditions Not concurrently on hypertransfusion program

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1997-11; Study Completion 1999-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Martin Emanuele, Study Chair — CytRx

REFERENCES:
- [Background] Adams-Graves P, Kedar A, Koshy M, Steinberg M, Veith R, Ward D, Crawford R, Edwards S, Bustrack J, Emanuele M. RheothRx (poloxamer 188) injection for the acute painful episode of sickle cell disease: a pilot study. Blood. 1997 Sep 1;90(5):2041-6. PMID 9292541